CLINICAL TRIAL: NCT07126691
Title: " Investıgatıon Of Changes In Flexıbılty And Lung Capacıty Among Gırls Begınner Synchroızed Swımmıng And Free Style Swımmıng Between The Ages Of 6-9.".
Brief Title: " ISynchroızed Swımmıng And Free Style Swımmıng
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Feyza Sule BADILLI HANTAL, Asst.Prof, Yeditepe University
Other Study IDs: yüzme
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Healthy Young Children
Keywords: Synchronized swimming, freestyle swimming, pulmonary function, FVC, FEV1, flexibility, sit and reach test, dry-land exercises

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational cohort study aimed to investigate the effects of swimming style on pulmonary function and flexibility in young female swimmers. A total of 24 beginner swimmers (12 synchronized swimmers and 12 freestyle swimmers; aged 6-9 years) from swimming clubs in Istanbul, Turkey, were evaluated between January and April 2019. Pulmonary function was assessed using spirometry, measuring Forced Vital Capacity (FVC) and Forced Expiratory Volume in 1 second (FEV1). Flexibility was assessed by the Sit and Reach test. Assessments were performed at baseline and after a 3-month training period. No statistically significant differences were found between the two groups in terms of changes in FVC, FEV1, or flexibility improvement (p > 0.05). However, both groups showed significant within-group improvements in flexibility over time. Longer-term studies with larger sample sizes may yield more conclusive results.

DETAILED DESCRIPTION:
This study evaluated the influence of swimming style and associated dry-land training on pulmonary function and flexibility in young female swimmers over a 3-month period. Participants were beginner synchronized swimmers and freestyle swimmers, aged 6-9 years, recruited from different swimming clubs in Istanbul, Turkey. Pulmonary function was measured using spirometry, including Forced Vital Capacity (FVC) and Forced Expiratory Volume in 1 second (FEV1). Flexibility was assessed by the Sit and Reach test. Both assessments were performed at the start and at the end of the study period. While no statistically significant between-group differences were detected for pulmonary parameters or the degree of flexibility improvement, both groups demonstrated significant within-group improvements in flexibility. The findings suggest that swimming training, regardless of style, may enhance flexibility in young athletes.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have no systemic health problems,between 6-9 ages beginner level girls and trains twice a week.The swimmers who met inclusion criteria are divided into two groups as synchronized swimmers (SG) and free style swimmers (FG) . Swimmers was selected from the groups that have just started swimming, ie those who have been swimming for max 2 months.

Exclusion Criteria:

* Children training more than twice a week and doing another sport or sports are excluded.

Ages: 6 Years to 9 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Beginner female synchronized swimmers and freestyle swimmers, aged 6 to 9 years, who were actively training in swimming clubs in Istanbul, Turkey. Participants had no known respiratory, cardiovascular, or musculoskeletal disorders and were able to perform standard pulmonary function and flexibility tests.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Forced Vital Capacity (FVC) - measured by spirometry at baseline and after 3 months. | (Time Frame: 3 months
  Change in Forced Vital Capacity (FVC) - Pulmonary function will be assessed using spirometry. FVC will be recorded in liters at baseline and after a 3-month training period to evaluate changes in lung capacity associated with swimming style. (Time Frame: 3 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided